CLINICAL TRIAL: NCT06621446
Title: The Beijing Adult Dry Eye Cohort Study
Acronym: ADEC
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Ying Jie, MD, Prof, Beijing Tongren Hospital
Other Study IDs: BeijingTH TREC2024-KY084; Xue Ke Dai Tou Ren-02-22 (Registry Identifier: Beijing Tongren Hospital); Xue Ke Dai Tou Ren-02-22 (Other: Beijing Tongren Hospital)
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye
Keywords: Prevalence; Incidence; Risk Factor; Dry Eye; Adult
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive intervention model — A dry eye intervention strategy: including health education, the use of eye drops, and regular review.

SUMMARY:
To investigate the prevalence of dry eye in adults in Beijing, and explore the extremely dangerous factors of dry eye in adults in Beijing through two years follow-up, and establish a prediction model of dry eye; On this basis, the prevention and treatment strategy of dry eye disease suitable for Chinese people is put forward, and its actual effect is verified.

DETAILED DESCRIPTION:
Specifically, it is planned to carry out cluster random sampling in Jianguomen community, Yongdingmenwai community, and Jiaodaokou community in Dongcheng District, Beijing, and select adults over the age of 18 to enter the queue for observation; In order to ensure the accuracy of the prevalence survey, people with mobility difficulties or mental problems are not excluded. The subjects will be examined by ophthalmology and OSDI questionnaire to determine whether these people have dry eyes. Then the prevalence of dry eye would be expolored. Then through one-year and two-year follow-up, the incidence would be explored.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above, resident population of sample community, able to complete dry eye examination, informed consent signed

Exclusion Criteria:

* Mental illness, mobility difficulties, can not participate in follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a population-based study. Study population are residents (adults aged above 18) of sampled communities.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dry eye | two years
  The incidence of dry eye is the primary outcome, and will be calculated by number of newly developed dry eye cases divided by total number of those who didn't have dry eye in last year.
  The presence of dry eye will be measured relying on the following examinations: questionnaire, tear break-up time examination

SECONDARY OUTCOMES:
Prevalence of Dry Eye | one year
  The prevalence of dry eye is the secondary outcome. The prevalence will be defined as number of dry eye cases, divided by total participants. Dry eye will be measured relying on questionnaire and tear break-up time examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided